CLINICAL TRIAL: NCT02028481
Title: Air Tamponade in Macular Holes < 400 μm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012815b1
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Macular Holes
Keywords: Macular hole; Vitreoretinal surgery; Macular surgery; Air tamponade
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Postoperative air tamponade (Experimental): Pars plana vitrectomy, ILM peeling and air tamponade. No postoperative face down positioning. All patients need to be pseudophakic prior to intervention.
  Interventions: Procedure: Postoperative air tamponade

INTERVENTIONS:
Procedure: Postoperative air tamponade — Pars plana vitrectomy, ILM peeling and air tamponade. No postoperative face down positioning. All patients need to be pseudophakic prior to intervention.

SUMMARY:
Macular hole is a hole formation which takes place in the center of the retina. Such a hole needs surgical steps in order to close. Closure of the macular hole will lead to a substantially improvement of vision in most cases. Following macular hole surgery a tamponade of intraocular gas is normally injected in order to keep the macula dry for the postoperative period. Postoperative face down position for a week was earlier standard. Several authors report of good closure rates with both air tamponade or lack of face down positioning. In this study standard pars plana vitrectomy with peeling of the internal limiting membrane (ILM) will be performed. The gas tamponade will be replaced by air. Postoperative face down positioning will not be used. Only macular holes less than 400 μm will be included.

ELIGIBILITY:
Inclusion Criteria:

* Primary macular hole less than 400 μm in diameter
* Duration of symptoms less than 36 months
* Informed consent

Exclusion Criteria:

* Previous vitreomacular surgery
* Myopia more than 6 diopters
* Ocular trauma
* Disease affecting visual function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Closure rate of macular hole | 1 month after enrollment

OTHER OUTCOMES:
Visual gain after 6 months of follow up | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Forsaa, MD, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Department of Ophthalmology, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No